CLINICAL TRIAL: NCT00344825
Title: Observational Study for Evaluation of Quality of Life in Patients Under Treatment for B-Chronic Lymphocytic Leukemia.
Brief Title: Vitalis Study - Observational Study on the Quality of Life in Patients Under Treatment for B-Chronic Lymphocytic Leukemia (B-CLL)
Status: Completed | Type: Observational
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme
Organization: Sanofi (Industry)
Other Study IDs: 306003
Record Dates: First submitted 2006-06-26; First posted 2006-06-27 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Leukemia, B-Cell, Chronic
Keywords: B- Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, B-Cell | interventions — Alemtuzumab; fludarabine phosphate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Alemtuzumab (MabCampath, BAY86-5045) and Fludarabine Phosphate (Fludara, BAY86-4864)

INTERVENTIONS:
Drug: Alemtuzumab (MabCampath, BAY86-5045) and Fludarabine Phosphate (Fludara, BAY86-4864) — Descriptive statistical methods applied for the whole study cohort and for subgroups according to QoL and the correlation of the following parameters: Age, Sex, Stage of disease, Time from first B-CLL diagnosis, number of previous B-CLL treatments, Reason of starting of the new B-CLL treatment (progression disease, relapse, no-response to the previous treatment, previous treatment toxicity), Therapeutic Regimen (Day Hospital, Hospital Admission, etc.), Type of Centre, B-CLL treatment lasting, Response to B-CLL treatment.
  QoL at baseline, Change in QoL over time evaluated using an analysis of Variance.

SUMMARY:
300 patients, starting a new pharmacological treatment for B-CLL, were enrolled by 36 Italian Centres for assessing the Quality of Life (QoL). A descriptive analysis of QoL and the correlation of the age, sex, stage of disease, Time from first B-CLL diagnosis, Number of previous B-CLL treatments, reason of starting of the new B-CLL treatment: therapeutic Regimen, type of Centre, B-CLL treatment lasting, response to B-CLL treatment.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.

Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Aged >/=18 years
* Patients of either sex with B-CLL, who are starting a new pharmacological treatment for B-Chronic Lymphocytic Leukemia (1st, 2nd, 3rd, 4th)
* Foreseen duration of CLL therapy </= 6 months
* B-Chronic Lymphocytic Leukemia progressive stage A, stage B or C (according to Binet system), or II-IV (according to Rai system)
* WHO Performance Status </= 2
* Life expectancy </= 6 months
* Signed Informed consent for personal data's treatment and availability to fill in the QoL questionnaire

Exclusion Criteria:

* Patients with any other tumour disease
* Chronic Lymphocytic Leukemia therapy in the last 30 days before V0
* More than 3 previous CLL treatments (the therapy is defined by the drug and/or the treatment period)
* Previous stem cells transplantation
* Concurrent or in the last 30 days participation to any other clinical trial
* Any medical or psychological conditions that might compromise the capacity to sign the consent for personal data's treatment or to fill in the QoL questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, aged >/= 18 years, either sex with B-CLL, who are starting a new pharmacological treatment for B-CLL (1st, 2nd, 3rd, 4th), duration of CLL therapy </= 6 months, WHO Performance Status ≤ 2, life expectancy >/= 6 months
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2004-01; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- Many Locations, Italy